CLINICAL TRIAL: NCT07301593
Title: Comparison of Two Ankle Foot Orthosis on Mobility, Participation and Adhesion in Childrend With Cerebral Palsy
Acronym: DynamicPC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DynamicPC; 2025-A00301-48 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
Keywords: orthosis-propulsion-running-children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group carbon/plastic (Active Comparator): crossover
  Interventions: Other: orthosis use
- Group A (Active Comparator): crossover
  Interventions: Other: orthosis use

INTERVENTIONS:
Other: orthosis use — Participants assigned to this group will wear the c-AFO for a 4-week intervention period. Outcome assessments will be conducted at baseline and at the end of the 4-week period. Following a 2-week washout phase, participants will then wear the pl- AFO for an additional 4 weeks, with identical outcome assessments performed at the corresponding baseline and endpointPlastic ankle foot orthosis or carbon ankle foot orthosis

SUMMARY:
Children with cerebral palsy (CP) present a variety of motor impairments and activity limitations. Plastic ankle-foot orthoses (pl-AFO) are frequently prescribed to improve their gait. However, their use limit forward propulsion generation, which explains why children tend to remove their pl-AFO during recreational activities,including running and jumping. While the benefits of physical activity are proven for these children, there is no data about pl-AFO impact across a range of locomotor activities. Biomechanically optimized dynamic carbon fiber AFOs (c-AFO) are now available and may improve propulsion features in comparison with usual pl-AFOs. The investigators aim to compare the AFO-specific effects (pl-AFO vs c-AFO) on propulsion (during walking, running and jumping), to explore the consequences on social participation, as well as to evaluate the effect on the hemiparetic CP child's perception and adherence of wearing each AFO. In this prospective, multicenter, randomized controlled trial with a crossover design, 38 hemiparetic CP children from 8 to 15 years old will be evaluated with their usual pl-AFO and with a c-AFO. The pragmatic clinical approach of this study is expected to provide data to guide and optimize AFO prescription and use, while enhancing understanding of these devices and their adaptation to the actual physical activity of CP children.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with a crossover design. A total of 38 patients will be recruited from three different centers.

Each participant will be randomly assigned to one of two groups (Group c/pl or Group pl/c). Depending on the group allocation, each subject will test both types of ankle-foot orthoses (AFOs) in a different order.

* Group c/pl: Participants in Group A will first use the carbon AFO (c-AFO) for four weeks. Evaluations will be conducted before and after this period. After a washout phase, they will then use the plastic AFO (pl-AFO) for another four weeks, with evaluations conducted before and after this second phase.
* Group pl/c: Participants in Group B will follow the same protocol, but in reverse order: starting with the pl-AFO for four weeks (with pre- and post-evaluations), followed by a washout period and then four weeks with the c-AFO (again with evaluations before and after).

Each evaluation includes:

* A quantitative gait analysis including ground reaction force measurements, kinematic data, and spatiotemporal parameters.
* Clinical tests to assess functional mobility and endurance.
* Questionnaires to evaluate participation levels, satisfaction, and acceptance of the AFOs.

ELIGIBILITY:
Inclusion Criteria:

* Children from 8 to 15 years old
* Spastic, hemiparetic cerebral palsy
* Level I or II on the Gross Motor Function Classification System
* Ability to walk and run 10 meters without assistance
* Ability to jump (simultaneous lift of both feet)
* Daily use of a plastic ankle foot orthosis allowing ankle mobility
* Affiliated to a social security scheme

Exclusion Criteria:

* Children with ataxic, dyskinetic, or mixed-type cerebral palsy
* Children with cognitive, intellectual, or behavioral disorders that may impair their understanding of instructions, the proper conduct of evaluations, or the use of assessment scales, as judged by the investigator.
* Children who have received botulinum toxin injections within 4 months prior to the inclusion visit
* Children or adolescents who have undergone surgical intervention:

within the past 6 months prior to inclusion if no bony procedure was performed, or within the past 12 months prior to inclusion if a bony procedure was performed, or who have a planned surgical procedure during the study period.

* Children who have participated in an intensive rehabilitation program within 4 months prior to the inclusion visit
* Children or adolescents participating in another interventional study that could interfere with the outcomes of the present study by altering the subject's physical abilities.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Propulsion force during running | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period.
  Anteroposterior component of the ground reaction force (GRF), recorded during running, using force plates

SECONDARY OUTCOMES:
force plates | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period.
  Propulsion forcesduring jumping and walking (force plates)
Quantitative gait analysis | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period.
  Kinematics parameters during running, jumping and walking
Quantitative Gait analysis | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period
  Spatiotemporal parameters during running, jumping and walking: Step length, foot clearance, single and double support time, flight phase duration during running and jump height.
Running endurance | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period.
  Running endurance (using the 10 Meters Shuttle Run Test)
Functional mobility | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period
  Items D and E of the Gross Motor Function Measure, with a total score ranging from 0 to 111.
Participation in physical activities | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period
  Participation in physical activities, using the Children and Adolescent Physical Activity and Sedentary Questionnaire. The questionnaire includes two subscales: physical activity, scored from 1 to 4, and sedentary behavior, scored from 1 to 6
Adhesion toward the AFOs | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period
  By a Follow up booklet
Tolerance toward the AFOs | At baseline and at the end of the intervention (4 weeks) for the 2 interventions period
  By a follow up booklet

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MEDERER, Principal Investigator — Hôpital Raymond Poincaré - Service Neurologie Pédiatrique Médecine Physique et Réadaptation
Locations (1):
- Hôpital Raymond Poincaré - Service Neurologie Pédiatrique Médecine Physique et Réadaptation, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided